CLINICAL TRIAL: NCT04968080
Title: Prospective, Observational, Single-Arm Study to Validate Comparability of an Infrared Thermographic Camera Versus Oral, Forehead, and Ear Thermometers When Determining Body Temperature in Anonymous Adult Participants
Brief Title: A Study to Validate Comparability of an Infrared Thermographic Camera Versus Oral, Forehead, and Ear Thermometers When Determining Body Temperature in Adult Participants
Status: Completed | Type: Observational
Sponsor: Infrared Cameras Incorporate (Industry)
Responsible Party: Sponsor
Other Study IDs: ICI IRT V 001
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Temperature Change, Body
Keywords: Infrared Thermal Camera; IRT
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Full Analysis Set: Participants will have their temperature collected by infrared thermal camera (IRT), oral, forehead, and ear thermometers.
  Interventions: Device: Infrared Cameras Inc. (ICI) FMX 400 Infrared (IR) Camera System; Device: Welch Allyn SureTemp Plus 690; Device: Welch Allyn ThermoScan PRO 6000; Device: Infrared Cameras Inc. (ICI) HotSpot Infrared (IR) NonContact Infrared Thermometer

INTERVENTIONS:
Device: Infrared Cameras Inc. (ICI) FMX 400 Infrared (IR) Camera System — Infrared thermal camera
Device: Welch Allyn SureTemp Plus 690 — Oral thermometer
Device: Welch Allyn ThermoScan PRO 6000 — Ear thermometer
Device: Infrared Cameras Inc. (ICI) HotSpot Infrared (IR) NonContact Infrared Thermometer — Forehead temperature gun

SUMMARY:
The primary objective of this study is to determine if the Infrared Cameras, Inc (ICI) FMX 400 infrared (IR) Class 1 infrared thermal camera (IRT) system is comparable to oral, forehead, and ear thermometers for determining human body temperature.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide opt-out consent.
2. Participants must agree to have temperature recorded noninvasively using an infrared thermal camera (IRT) Class 1 device, oral thermometer, forehead thermometer, and ear thermometer.

Exclusion Criteria:

1. Participants who opt out of participating; ie, participants who do not agree to have temperature recorded noninvasively using an IRT Class 1 device, oral thermometer, forehead thermometer, and ear thermometer.
2. Participants who are not able to understand that their temperature will be recorded, or who are otherwise unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants entering the PRA Health Sciences - Early Development Services (PRA-EDS) Salt Lake City business location who agree to receive anonymous infrared thermal camera (IRT) Class 1 device temperature scan while undergoing routine temperature surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Infrared Thermal Camera (IRT) Calculated Human Body Temperature | Up to Week 4
Average Oral Thermometer Body Temperature | Up to Week 4
Forehead Thermometer Body Temperature | Up to Week 4
Average Ear Thermometer Body Temperature | Up to Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences - Early Development Services, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No